CLINICAL TRIAL: NCT06903715
Title: An Open-Label, Phase 1 Study to Characterize the Effects of Phenytoin on the Pharmacokinetics of Belzutifan in Healthy Adult Participants
Brief Title: A Clinical Study of Belzutifan (MK-6482) Alone or With Phenytoin in Healthy Participants (CA46602/MK-6482-035)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 6482-035; CA46602 (Other: Celerion)
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Healthy
MeSH Terms: interventions — belzutifan; Phenytoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Belzutifan + Phenytoin (Experimental): Participants receive belzutifan during study Period 1, followed by a washout period, then they receive belzutifan and phenytoin during study Period 2.
  Interventions: Drug: Belzutifan; Drug: Phenytoin

INTERVENTIONS:
Drug: Belzutifan — Oral administration
  Other Names: MK-6482; PT2977; Welireg™
Drug: Phenytoin — Oral administration
  Other Names: Phenytoin sodium

SUMMARY:
Researchers designed belzutifan, the study medicine, to treat certain kinds of cancer.

The goal of this study is to learn what happens to belzutifan in a healthy person's body over time when taken, by mouth, as a tablet. Researchers will learn what happens when belzutifan is taken alone and when it is taken after several days of treatment with phenytoin.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Healthy, adult, male (vasectomized or surgically sterilized) or female (of non-childbearing potential)
* Has a body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the participant by their participation in the study
* History or presence of: Seizure (excluding simple febrile seizure), epilepsy, severe head injury, multiple sclerosis, or other known neurological conditions which the PI considers to be clinically significant; Hypersensitivity reaction to anticonvulsant therapy (including phenytoin, primidone, and phenobarbital); Depression, unusual changes in mood or behavior or suicidal thoughts and behavior; Hepatic porphyria (e.g., acute intermittent porphyria, variegate porphyria, porphyria cutanea tarda)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2025-03-28 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of Belzutifan | Predose and at designated timepoints up to 120 hours postdose
  Blood samples will be collected to determine the AUC0-inf of belzutifan.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 36 days
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Drug Due to an AE | Up to approximately 22 days
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study due to an AE will be reported.
Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-last) of Belzutifan in Plasma | Predose and at designated timepoints up to 120 hours postdose
  Blood samples will be collected to determine the AUC0-last of belzutifan.
Area Under the Concentration-Time Curve from Time 0 to 24 Hours (AUC0-24) of Belzutifan in Plasma | Predose and at designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the AUC0-24 of belzutifan.
Maximum Plasma Concentration (Cmax) of Belzutifan in Plasma | Predose and at designated timepoints up to 120 hours postdose
  Blood samples will be collected to determine the Cmax of belzutifan.
Plasma Concentration 24 Hours Postdose (C24) of Belzutifan in Plasma | 24 hours postdose
  Blood samples will be collected to determine the C24 of belzutifan.
Time to Maximum Plasma Concentration (Tmax) of Belzutifan in Plasma | Predose and at designated timepoints up to 120 hours postdose
  Blood samples will be collected to determine the Tmax of belzutifan.
Apparent Terminal Half-life (t1/2) of Belzutifan in Plasma | Predose and at designated timepoints up to 120 hours postdose
  Blood samples will be collected to determine the t1/2 of belzutifan.
Apparent Clearance (CL/F) of Belzutifan in Plasma | Predose and at designated timepoints up to 120 hours postdose
  Blood samples will be collected to determine the CL/F of belzutifan.
Apparent Volume of Distribution during terminal phase (Vz/F) of Belzutifan in Plasma | Predose and at designated timepoints up to 120 hours postdose
  Blood samples will be collected to determine the Vz/F of belzutifan.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion, Inc. ( Site 0001), Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/